CLINICAL TRIAL: NCT04991090
Title: Management of Clinically Involved Lateral Lymph Node Metastasis in Locally Advanced Rectal Cancer: A Prospective Radiation Dose Escalation Study
Brief Title: Management of LLN Metastasis in Locally Advanced Rectal Cancer: A Prospective Radiation Dose Escalation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dose-esclation-LLN
Record Dates: First submitted 2021-05-26; First posted 2021-08-05 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: dose escalation of lymph node metastasis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- escalation (Experimental): The gross tumor volume (GTV) was defined as gross disease determined on MRI scans. The clinical target volume (CTV) was defined as the GTV plus areas considered at significant risk of harboring microscopic area. The lymph nodes (SA ≥ 5 mm) existed at the internal iliac and obturator would be delineated, named as GTVnd, and received a radiation dose boost. The planning target volume (PTV) was generated by adding an 8-mm margin around the GTV, GTVnd, and CTV in all directions. Doses of 58 Gy, 50 Gy, and 45 Gy were delivered to PTV-GTVnd, PTV-GTV, and PTV-CTV at 25 fractions, respectively. The dose of the normal organs at risk was constrained to the following criteria: bowel bag, V50 ≤ 5%; bladder, V50 ≤ 50%; femoral heads, V50 ≤ 5% .
  Interventions: Radiation: escalation dose of LLNs

INTERVENTIONS:
Radiation: escalation dose of LLNs — The lymph nodes (SA ≥ 5 mm) existed at the internal iliac and obturator would be delineated, named as GTVnd, and received a radiation dose boost of 58Gy.
  Other Names: escalation group

SUMMARY:
In this study, locally advanced rectal cancer (LARC) patients with lateral lymph node (LLN) metastasis would be enrolled. The LLNs with short axis (SA) ≥ 5 mm are considered metastatic.The safety of neoadjuvant chemoradiotherapy(nCRT) with a booster dose to 58Gy had been initially demonstrated in our previous research. The effective and safety of dose escalation of LLN in LARC patients, will be further verified in this prospective, clinical study.

DETAILED DESCRIPTION:
This is a prospective, observational clinical study for validation the efficiency and safety of the dose escalation of LLN. Patients who have been pathologically diagnosed as rectal adenocarcinoma and defined as clinical T1-4N1-2M0 without distant metastasis will be enrolled from the Sixth Affiliated Hospital of Sun Yat-sen University. Patients should have at least one LLN metastasis defined on primary MRI, and the data of primary pelvic MRI will be performed within two weeks before the beginning of enrollment. All patients should follow a standard treatment protocol, including concurrent neoadjuvant chemoradiotherapy (nCRT) with a dose boost of LLNs to 58Gy, TME surgery with or without LLND ( lateral lymph node dissection) and adjuvant chemotherapy. The regimen of chemotherapy and the way of operation should be depended on the MDT(multiply discipline treatment) decision. The restaged MRI scan would be performed 6-12 weeks after the last fraction of radiotherapy. The LLN response rate ( short axis < 5mm ) would be evaluated. This study is aimed to apply a new way to control LLN metastasis.

ELIGIBILITY:
Inclusion Criteria:

* informed consent was signed ;
* Age 18-75;
* Pathologically confirmed rectal adenocarcinoma, colonoscopy,MRI, CT and other examinations confirmed that the tumor was located under peritoneal reflexion,
* clinical staging was T1-4N1-2M0, pelvic MRI evaluation showed at least one lateral lymph node with short diameter ≥5 mm;
* Pelvic MRI was evaluated no more than 14 days before enrollment;
* ECOG 0-2 points;
* No prior history of other malignant tumors, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Exclusion Criteria:

* Previous radiotherapy or surgical treatment for colorectal cancer (except biopsy for pathology);
* Whole body CT, MR or PET-CT (including at least chest, whole abdomen, and pelvis) confirmed distant metastasis (M1);
* Previous or coexisting active malignancies (other than malignant neoplasms that have received curable treatment and have not been present for more than 3 years or carcinoma in situ that can be cured by adequate treatment);
* Receiving major operations such as laparotomy, thoracotomy, laparoscopic resection of organs or serious external injuries within the previous 4 weeks;
* Active coronary artery disease, severe/unstable angina pectoris or newly diagnosed angina or myocardial infarction within the 12 months prior to study participation;
* Patients who have experienced thrombosis or embolism within the past 6 months have received radiotherapy or surgical treatment for rectal cancer (except biopsy for pathology)
* New York Heart Society (NYHA) Grade II or higher congestive heart failure;
* The presence of CTCAE grade 2 or above toxicity (except anemia, alopecia, and skin pigmentation) due to any previous treatment that has not resolved;
* Pregnant or lactating women;
* Accompany with any medical condition that would affect patient safety and study compliance;
* Patients determined by the investigator to be unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
the responsive rate of dose escalation of LLN | 3 years
  the LLN responsive rate (short diameter < 5mm) of neoadjuvant chemoradiotherapy combined with dose escalation of LLN in the treatment of middle and low locally advanced rectal cancer

SECONDARY OUTCOMES:
prognosis outcome-3-year Local Recurrence | 3 years
  The 3-year Local Recurrence of LARC patients underwent neoadjuvant chemoradiotherapy combined with dose escalation of LLN
prognosis outcome-3-year Lateral Local Recurrence | 3 years
  The 3-year Lateral Local Recurrence of LARC patients underwent neoadjuvant chemoradiotherapy combined with dose escalation of LLN

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbo Wan, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China